CLINICAL TRIAL: NCT00172081
Title: An 18-Month Double-Blind, Placebo-Controlled, Phase III, Trial With a 12-Month Interim Analysis of the Effect of Recombinant Human Parathyroid Hormone (ALX1-11) on Fracture Incidence in Women With Postmenopausal Osteoporosis
Brief Title: TOP: Recombinant Human Parathyroid Hormone (ALX1-11) on Fracture Incidence in Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALX1-11-93001
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Osteoporosis
Keywords: Post-menopausal; Osteoporosis; Parathyroid Hormone; PTH; ALX1-11
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Daily subcutaneous injection into thigh or abdomen with 700 mg Calcium and 400 IU Vitamin D daily
  Interventions: Drug: placebo
- PTH(1-84) 100 mcg (Experimental): Subcutaneous injection of PTH(1-84) with 700 mg Calcium and 400 IU Vitamin D daily
  Interventions: Drug: ALX1-11

INTERVENTIONS:
Drug: placebo — Daily subcutaneous injection with placebo
  Arms: placebo
Drug: ALX1-11 — PTH (1-84) 100 mcg injected subcutaneously into the thigh or abdomen
  Other Names: PREOS
  Arms: PTH(1-84) 100 mcg

SUMMARY:
This is an 18-month, double-blind, placebo-controlled, Phase III trial with a 12-month interim analysis of the effect of ALX1-11, recombinant human parathyroid hormone (1-84) (rhPTH [1-84]), on fracture incidence in women with postmenopausal osteoporosis, the TOP study.

DETAILED DESCRIPTION:
Parathyroid hormone (PTH), a polypeptide consisting of 84 amino acids that is synthesized and secreted by the parathyroid glands, is a principal regulator of calcium homeostasis through concerted action on kidney, intestine and bone. Parathyroid hormone exerts its action on bone to release calcium into the extracellular fluid as a process of bone remodeling and also to maintain the serum calcium concentration, but the exact mechanisms are not fully understood. In some circumstances, PTH may exert an anabolic action on bone and can stimulate osteoblast proliferation and mature osteoblast function. The net effect of exogenous PTH administration on bone turnover depends on the pattern of delivery. A continuous long-term infusion gives a net decrease in trabecular bone volume, whereas daily single injections result in a net increase.

NPS Allelix Corp. is developing ALX1-11, recombinant human parathyroid hormone (1-84), for the treatment of osteoporosis. ALX1-11 is identical to the endogenous intact 84 amino acid human hormone and will be self-administered on a daily basis by subcutaneous (sc) injection.

Currently, there is no approved therapy for osteoporosis capable of stimulating the formation of new bone of normal composition and structure. Most therapies in development are anti-catabolic and only prevent further bone loss (e.g., estrogen replacement, bisphosphonates, and calcitonins). ALX1-11 has the potential to stimulate new bone formation in osteoporotic patients, thereby increasing bone mass and preventing fractures. Patients with moderately or severely reduced bone density and a fracture would be expected to benefit from treatment, thereby improving functional status and alleviating symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women who are postmenopausal with at least one year since the last menstruation.
* Women who are 45-54 years of age with the following bone mineral density (BMD) and/or vertebral fracture:

  * BMD 3.0 standard deviations (SDs) or more below peak bone mass of young females at the lumbar spine, femoral neck, or total hip; or
  * BMD 2.5 SDs or more below peak bone mass of young females at the lumbar spine, femoral neck or total hip with the presence of a vertebral fracture verified by the central imaging organization before the patient is enrolled into the study.
* Women 55 or more years of age with the following BMD and/or vertebral fracture:

  * BMD 2.5 SDs or more below peak bone mass of young females at the lumbar spine, femoral neck or total hip; or
  * BMD 2.0 SDs or more below peak bone mass of young females at the lumbar spine, femoral neck or total hip with the presence of a vertebral fracture verified by the central imaging organization before the patient is enrolled into the study.
* The following types of vertebral fractures should not be considered for patient enrollment into this trial:

  * Pathological fractures due to malignant disease or infection
  * Fractures due to excessive trauma sufficient to cause a fracture in young individuals with normal bone mass
* Women with the ability to self-administer a daily injection or have a designee who will give the injections
* Women who are capable of understanding and giving written, voluntary informed consent before the clinical trial screening visit

Exclusion Criteria:

A. Vertebral Deformity:

* Patient has 5 or more vertebral (thoracic and lumbar) deformities
* Patient has 2 or more lumbar vertebral deformities (L1 to L4)
* Severe lumbar scoliosis (>15 degrees) which precludes a reliable evaluation of the dual x-ray absorptiometry (DXA)

B. DXA Imaging:

* Inability to have a DXA scan performed.

C. History or Concurrent Illness:

* Disorders of immunity
* Endocrine system
* Gastrointestinal system
* Kidney and collecting system
* Liver, biliary tract and pancreatic systems
* Musculoskeletal system
* Neoplasia
* Nervous system
* Vascular, respiratory and cardiac system
* Significant diseases or disorders are determined by history, physical exam or laboratory screens and judged by the Principal Investigator to be significant.

D. Concurrent Medication:

Any patient who does not require medication washout (discontinuation) as specified below may start study drug dosing after 2 weeks of stabilization treatment with calcium and vitamin D3 supplements. All exceptions will be documented in the case report form (CRF).

* Patients cannot be enrolled into this clinical trial if they have received any of the following therapies at any time:

  * Any PTH or PTH analogs [e.g., rhPTH(1-84), PTH(1-34), PTHrP and analogs]
  * Fluoride
  * Strontium
* Patients must have been off the following agents for the specified times before entering the screening phase of this clinical trial:

  * Any investigational drug (30 days)
  * Anabolic steroids or androgens (6 consecutive months)
  * Active vitamin D3 metabolites and analogs(90 days)
  * Systemic corticosteroids, more than 5 mg/day prednisone or a systemic corticosteroid formulation equivalent to 5 mg/day prednisone (12 consecutive months).
  * A patient who has been enrolled in the study and needs to receive an acute bolus of steroids (oral or injectable) for a self-limited illness may continue treatment in the study if the following requirements are met:

    1. Exposure to steroids is limited to no more than 30 consecutive days
    2. The maximal dose of steroid (prednisone equivalent) is limited to no more than 225 mg (7.5 mg each day for 30 days)
    3. The illness is acute in nature and is not expected to recur during the remaining treatment period of the study
  * Daily inhaled corticosteroids unless dose is below 1200 mg/day of beclomethasone.
  * Bisphosphonates, including investigational bisphosphonates.
  * Intravenous (IV) pamidronate. Patient must be receiving pamidronate specifically to treat osteoporosis. Patient can have received only ONE IV dose of pamidronate in the 12 months immediately preceding the screening visit.
  * Cyclical etidronate. Exposure to cyclical etidronate must be less than or equal to 6 months on a standard dose (e.g. 400 mg/day). Patient should not have exposure to cyclical etidronate for 9 months prior to the screening visit.
  * Phenytoin for seizure control. If the patient has received phenytoin within five years of the screening visit, the patient is excluded from this study. The patient may continue in the screening process if 15 years have passed since the last dose of phenytoin at the time of the screening visit. If the phenytoin use was between 5-15 years before the screening visit and the patient received phenytoin for less than 2 months.
* Patients may be enrolled if they have been stabilized on the following therapy for the specified amount of time:

  * Thyroid hormone (<0.1 mg/day thyroxine) therapy for at least 6 months. * Stable dosage of thiazide for at least 3 consecutive months.
* All patients must stop the following therapies at least 4 weeks prior to the screening visit and remain off these therapies for the remainder of the clinical trial. Screening laboratories must be performed after the washout is complete. However, imaging studies (BMD, X-rays) may be performed prior to starting the calcitonin, estrogen, and selective estrogen receptor modulation (SERM) washout.

  * Calcitonin
  * Estrogen replacement therapy by oral, transdermal or intramuscular administration
  * SERM drugs, e.g., tamoxifen, raloxifene, Evista
  * Vaginal application of estrogen-containing creams unless the dose is conjugated estrogen or estradiol* Cytostatics, e.g., azathioprine, recombinant human tumor necrosis fusion (Fc) protein, monoclonal antibody against tumor necrosis factor (e.g., remicade [infliximab])
  * The drug class tetracyclines
  * Medication known to affect the metabolism of bone (the Principal Investigator should discuss this with the Project Medical Officer before the patient is excluded from enrollment)

E. Miscellaneous Concurrent Medications:

* Methotrexate
* Intra-articular injections - Patients with chronic, active joint disease should be excluded from this Phase III study. Patients may receive a maximum of one intra-articular injection (ONE JOINT ONLY) every 6 months while participating in this Phase III study. The dose of corticosteroid injected should not exceed the anti-inflammatory equivalent dose of prednisone 40 mg suspension. The dose and volume should be adjusted downward as appropriate to the size of the joint.
* Provera is an acceptable concomitant medication when used according to the label instructions.

F. Laboratory Values and Physical Examination Findings:

* Serum calcium greater than 10.7 mg/dL (2.66 mmol/L). At screening, if the serum calcium is abnormal, the patient may have the additional evaluation described below ONCE:

  1. Discontinue all oral calcium and vitamin D3 supplements.
  2. Repeat a fasting serum calcium level two weeks later.
  3. If the fasting serum calcium level is still abnormal, the patient is discontinued from the study.
  4. If the repeat fasting serum calcium is normal, the patient should have supplemental calcium and vitamin D3 restarted at the time of study drug dosing, without going through a two-week stabilization period.
* Serum creatinine > 1.5 mg/dL (132.6 mmol/L)
* Urinary calcium to creatinine ratio is greater than or equal to 1. At screening, if a patient's urinary calcium to creatinine ratio is abnormal, the patient may have the additional evaluation described below ONCE:

  1. Discontinue all oral calcium and vitamin D3 supplements.
  2. Repeat a fasting urine calcium to creatinine ratio two weeks later.
  3. If the fasting urinary calcium to creatinine ratio is still abnormal, the patient is discontinued from the study.
  4. If the repeat fasting urinary calcium to creatinine ratio is normal, the patient should have supplemental calcium and vitamin D3 restarted at the time of study drug dosing, without going through a two-week stabilization period.
* Total serum alkaline phosphatase >130 U/L except as noted - Argentina (311 U/L); Brazil (278 U/L); Mexico (159 U/L).
* Any other clinically significant abnormal value as judged by the investigator
* Body weight below 40 kg

G. Substance Abuse:

* Alcohol and/or drug abuse

H. Psychiatric Disease:

* Current or history of psychiatric disease that would interfere with the ability to comply with the clinical trial protocol

I. Compliance:

* Suspected or confirmed poor compliance in completing clinical trial evaluations and/or clinical trial required questionnaires

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2532 (Actual)
Dates: Start 2000-04-27 (Actual); Primary Completion 2003-11-07 (Actual); Study Completion 2003-11-07 (Actual)

PRIMARY OUTCOMES:
Compare effects of 18 months of treatment with ALX1-11/placebo on the incidence of new and/or worsened thoracic and lumbar vertebral fractures in postmenopausal women with osteoporosis receiving calcium and vitamin D3 supplements | At Month 18

SECONDARY OUTCOMES:
Incidences of vertebral fractures at Month 12; hip and wrist fractures; and other clinical fractures. | At Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (174):
- United States (107):
  - Capstone Clinical Trials, Birmingham, Alabama
  - 'The University of Alabama at Birmingham, Birmingham, Alabama
  - 'Rheumatology Associates of North Alabama, Huntsville, Alabama
  - 'Radiant Research - Phoenix, Phoenix, Arizona
  - 'Robin K. Dore, M.D., Inc., Anaheim, California
  - 'Osteoporosis Medical Center, Beverly Hills, California
  - 'East Bay Clinical Trial Center, Concord, California
  - 'Loma Linda Osteoporosis Research Center, Loma Linda, California
  - 'The Foundation for Osteoporosis Research and Education, Oakland, California
  - 'Desert Medical Advances, Palm Desert, California
  - 'VA Palo Alto Health Care System, Palo Alto, California
  - 'Boling Clinical Trials, Rancho Cucamonga, California
  - 'Radiant Research - San Diego, San Diego, California
  - 'S.D. Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - 'San Francisco General Hospital, San Francisco, California
  - 'Community Research Centers, Santa Ana, California
  - 'Denver Arthritis Clinic, Denver, Colorado
  - 'Colorado Center for Bone Research, Lakewood, Colorado
  - 'Longmont Medical Research Network, Longmont, Colorado
  - 'Northeast Clinical Research, LLC, Hamden, Connecticut
  - 'Georgetown University Medical Center, Washington D.C., District of Columbia
  - 'RASF - Clinical Research Center, Boca Raton, Florida
  - 'ICSL Clinical Studies, Fort Myers, Florida
  - 'The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - 'Florida Wellcare Alliance, Inverness, Florida
  - 'Radiant Research - Lake Worth, Lake Worth, Florida
  - 'Osteoporosis Center University of Miami, Miami, Florida
  - 'Renstar Medical Group, Ocala, Florida
  - 'Diabetes and Endocrinology Treatment Center, Palm Beach Gardens, Florida
  - 'The Arthritis Center, Palm Harbor, Florida
  - 'The Centre for Arthritis and Rheumatic Diseases, South Miami, Florida
  - 'ICSL Clinical Studies, St. Petersburg, Florida
  - 'Radiant Research - Stuart & LakeWorth, Stuart, Florida
  - 'Palm Beach Research Center, West Palm Beach, Florida
  - 'The Emory Clinic, Atlanta, Georgia
  - 'Radiant Research, Honolulu, Hawaii
  - 'Intermountain Orthopaedics, Boise, Idaho
  - 'ICSL-Clinical Studies, Bloomington, Illinois
  - Rush-Prebyterian-St.Luke's Medical Center, Chicago, Illinois
  - 'The University of Chicago, Chicago, Illinois
  - 'University Hospital & Outpatient Center, Indianapolis, Indiana
  - 'Mercy Arthritis and Osteoporosis Center, Des Moines, Iowa
  - 'Wichita Clinic, Wichita, Kansas
  - 'Ochsner Clinic, New Orleans, Louisiana
  - 'Maine Center for Osteoporosis Research & Education, Bangor, Maine
  - 'Bethesda Health Research Center, Bethesda, Maryland
  - 'The Osteoporosis and Clinical Trials Center, Cumberland, Maryland
  - 'Arthritis & Osteoporosis Center of Maryland, Frederick, Maryland
  - 'The Osteoporosis and Clinical Trials Center, Hagerstown, Maryland
  - 'The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - 'Brigham & Women's Hospital, Boston, Massachusetts
  - 'Phase III Clinical Research, Fall River, Massachusetts
  - 'Osteoporosis Research & Treatment Center, Worcester, Massachusetts
  - 'Michigan Bone & Mineral Clinic, Detroit, Michigan
  - 'Desoto Family Medical Center, Olive Branch, Mississippi
  - 'St. John's Medical Research Group, Springfield, Missouri
  - 'VA Southern NV Healthcare Systems, Las Vegas, Nevada
  - 'Arthritis, Osteoporosis Muscle Skeletal Disease Center, Concord, New Hampshire
  - 'Comprehensive Clinical Research, Berlin, New Jersey
  - 'Anderson and Collins Clinical Research Inc., South Plainfield, New Jersey
  - 'New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - 'Lovelace Scientific Resources, Albuquerque, New Mexico
  - 'Bone Mineral Research Center, Mineola, New York
  - 'Beth Israël Medical Center, New York, New York
  - 'College of Physicians and Surgeons, Columbia University, New York, New York
  - 'Rochester Clinical Research Inc., Rochester, New York
  - 'Stony Brook Clinical Research Trials Center, Stony Brook, New York
  - 'Physicians Clinical Research Services, White Plains, New York
  - 'Carolina Bone and Joint - Charlotte, Charlotte, North Carolina
  - 'Duke University Medical Center, Durham, North Carolina
  - 'Odyssey Research Services, Bismarck, North Dakota
  - Michael J. Lillestol, Fargo, North Dakota
  - 'Altru Health Systems/Altru Research Center, Grand Forks, North Dakota
  - 'Odyssey Research Services, Minot, North Dakota
  - 'Cleveland Clinic Foundation, Cleveland, Ohio
  - 'David R. Mandel M.D. Inc., Mayfield, Ohio
  - 'Oklahoma Center for Arthritis Therapy & Research, Inc., Tulsa, Oklahoma
  - 'Osteoporosis Center, Medford, Oregon
  - 'Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - 'Thomas Jefferson University, Philadelphia, Pennsylvania
  - 'University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - 'Clinical Research Center of Reading LLP, West Reading, Pennsylvania
  - 'Radiant Research, Wyomissing, Pennsylvania
  - 'Rhode Island Hospital, Providence, Rhode Island
  - 'Roger Williams Medical Center, Providence, Rhode Island
  - 'Radiant Research, Anderson, South Carolina
  - 'Columbia Arthritis Center, PA, Columbia, South Carolina
  - 'Radiant Research, Greer, South Carolina
  - 'Rapid City Medical Center, Rapid City, South Dakota
  - 'Averna Research Institute, Sioux Falls, South Dakota
  - 'Brown Clinic, Watertown, South Dakota
  - 'Clinsearch, Chattanooga, Tennessee
  - 'Radiant Research/Dallas, Dallas, Texas
  - 'Breco Research Inc., Houston, Texas
  - 'Diabetes Center of the Southwest, Midland, Texas
  - 'Diabetes & Glandular Disease Research Associates, P.A., San Antonio, Texas
  - 'Radiant Research San Antonio, San Antonio, Texas
  - 'Salt Lake Women's Center, Sandy City, Utah
  - 'Fletcher Allan Health Center, UHC Campus 1, Burlington, Vermont
  - 'Center for Arthritis and Diabetes, Newport News, Virginia
  - 'National Clinical Research, Inc., Richmond, Virginia
  - 'MCV Physicians Program for Osteoporosis, Richmond, Virginia
  - 'South Puget Sound Clinical Research Center, Olympia, Washington
  - Phillip J. Mease, Seattle, Washington
  - 'Osteoporosis Research Group, Seattle, Washington
  - 'University of Wisconsin Medical Foundation, Madison, Wisconsin
  - 'Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (4):
  - 'IDIM, Buenos Aires, BUE
  - 'Centro Médico T.I.E.M.P.O, Buenos Aires, BUE
  - 'Hospital Ramos Mejía, Buenos Aires, BUE
  - 'Centro de Osteopatias Medicas, Capital Federal, CBA
- Brazil (10):
  - 'Universidade Federal do Paraná, Curitiba, Paraná
  - 'Universidade Federal de Pernambuco, Recife, Pernambuco
  - 'Hospital Santa Casa de Misericórdia do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - 'Hospital do Servidor Público do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - 'UNICAMP, Campinas, São Paulo
  - 'Pontifícia Universidade Católica de Campinas, Campinas, São Paulo
  - 'Hospital Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo
  - 'Universidade Federal de São Paulo, São Paulo, São Paulo
  - 'Instituto de Saúde e Bem Estar da Mulher, São Paulo, São Paulo
  - 'Hospital Heliópolis, São Paulo, São Paulo
- Bulgaria (5):
  - 'Multifunctional Hospital for Active Treatment "Sv.Georgy", Plovdiv
  - 'SHATENG"Acad.Ivan Penchev", Sofia
  - 'Multifunctional Hospital for Active Treatment "Alexandrovska, Sofia
  - 'Multifunctional Hospital for Active Treatment "Sv.Ivan Rilsky", Sofia
  - 'SHATGO"Sheynovo", Sofia
- Canada (22):
  - 'Heritage Medical Research Clinic, Calgary, Alberta
  - Osteoporosis Research Center, Vancouver, British Columbia
  - 'Manitoba Clinic, Winnipeg, Manitoba
  - Charlton Medical Centre, Hamilton, Ontario
  - Rafat Faraawi, Kitchener, Ontario
  - 'Centre for Activity and Aging, London, Ontario
  - St. Joseph's Health Centre, London, Ontario
  - 'Royal Victoria Hospital, Montreal, Ontario
  - Oakville Bone Center, Oakville, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - 'Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - 'St. Michael's Hospital, Toronto, Ontario
  - 'Osteoporosis Research Program, Toronto, Ontario
  - Jude F. Rodrigues, Windsor, Ontario
  - 'Riverside Medical Centre, Charlottetown, Prince Edward Island
  - 'Complexe Hospitalier de la Sagami, Chicoutimi, Quebec
  - 'Centre d'Etude Clinique Montreal Inc., Montreal, Quebec
  - 'Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - 'Centre de Recherche du CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Centre de Recherche - CORQ, Sainte-Foy, Quebec
  - Novabyss Research Clinic, Sherbrooke, Quebec
  - 'Saskatoon Osteoporosis Centre, Saskatoon, Saskatchewan
- Israel (9):
  - 'Soroka Medical Center, Beersheba
  - 'Clalit Health Services, Beersheba
  - 'Hillel Yaffe Medical Center, Hadera
  - 'Rambam Medical Center, Haifa
  - 'Lin Medical Center, Haifa
  - 'Hadassah University Hospital, Jerusalem
  - 'Rabin Medical Center, Petah Tikva
  - 'Chaim Sheba Medical Center, Ramat Gan
  - 'Lis Maternity Hospital, Tel Aviv
- Mexico (11):
  - 'Hospital Clinical del Parque, Chihuahua City, CHIH
  - 'Hospital Angeles de las Lomas, Huixquilucan, EMEX
  - 'Hospital Aranda de la Parra, León, Guanajuato
  - 'OPD Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - 'Hospital Civil de Belem, Guadalajara, Jalisco
  - 'Medica Monraz, Guadalajara, Jalisco
  - 'Osteosol, Mexico City, Mexico City
  - 'Instituto Mexicano de Investigacion Clinica, Mexico City, Mexico City
  - 'Hospital de Mexico, Mexico City, Mexico City
  - 'Hospital Central "Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí
  - 'Hospital Universitario de Monterrey, Monterrey Nuevo Leon
- Romania (3):
  - 'CLINTRIAL "DORIS" Medical Centre, Bucharest
  - 'Centrul Medical Sabyc, Bucharest
  - 'Spitalul Clinic Judetean Cluj-Napoca, Cluj-Napoca
- Russia (3):
  - 'Scientific Center of Endocrinology of RAMS, Moscow
  - 'JK "Medicine", Moscow
  - 'Russian Academy for Advanced Medical Studies, Moscow

REFERENCES:
- [Derived] Greenspan SL, Bone HG, Ettinger MP, Hanley DA, Lindsay R, Zanchetta JR, Blosch CM, Mathisen AL, Morris SA, Marriott TB; Treatment of Osteoporosis with Parathyroid Hormone Study Group. Effect of recombinant human parathyroid hormone (1-84) on vertebral fracture and bone mineral density in postmenopausal women with osteoporosis: a randomized trial. Ann Intern Med. 2007 Mar 6;146(5):326-39. doi: 10.7326/0003-4819-146-5-200703060-00005. PMID 17339618